CLINICAL TRIAL: NCT05918731
Title: Self-management in Chronic Obstructive Pulmonary Disease (COPD) Patients: A Primary Healthcare Intervention Study
Brief Title: Self-management in Chronic Obstructive Pulmonary Disease (COPD) Patients Compared to Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Izolde Bouloukaki, Principal Investigator, University of Crete
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: COPDSELF-1
Record Dates: First submitted 2023-05-24; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Self-Management

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (No Intervention): Patients who were assigned to receive usual care were instructed to continue up with their regular medical appointments and their usual check-ups/reviews and if they had any questions, to call the health coach.
- Self-management Intervention Group (Active Comparator): In the intervention group, a self-management program was implemented.
  Interventions: Behavioral: Self Management

INTERVENTIONS:
Behavioral: Self Management — A "training book" was given to this group, which was created for the study. The implementation process followed a five-step approach including sessions once a month for five consecutive months with a coach and follow-up phone calls after the end of the sessions.To inspire and engage patients, the sessions included a variety of educational techniques, including knowledge transfer, discussion, hands-on training, and homework. Additionally, coaches received training in motivational interviewing methods. The self-management program and all the process of data collection is described in detail on the supplementary file.
  Arms: Self-management Intervention Group

SUMMARY:
Evaluation of the effectiveness of COPD self-management interventions compared to usual on Quality of life, functional status, patient education, depression, and anxiety in primary healthcare users in the prefecture of Heraklion, Greece.

DETAILED DESCRIPTION:
To the best of our knowledge, no previous study has examined the effects of self-management programs on patients with COPD in Greece. Therefore, the investigators conducted a randomized controlled trial with a post-test design, to evaluate the implementation and clinical effectiveness of a COPD self-management intervention compared to usual care in terms of the following outcomes: Quality of life, functional status, patient education, depression, and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥18 years
* had previously been given a physician-diagnosis of mild COPD
* stable on their medications (no treatment modifications) in the last three months
* able to speak, read and/or understand Greek

Exclusion Criteria:

* refusal to participate
* concurrent oncological diseases
* severe cognitive impairment
* neurological, or psychiatric disability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Assessement of Quality of life | 6 months
  Assessment of the potential effect of self-management intervention on Quality of life using Short-Form Health survey (SF-12) questionnaire. The SF-12 is one of the most widely used instruments for assessing self-reported health-related quality of life. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Assessment of Functional status | 6 months
  Assessment of the potential effect of self-management intervention on functional status using COPD Clinical Questionnaire (CCQ) for clinically evaluating COPD.The Clinical COPD Questionnaire (CCQ) measures health status and can be used to assess health-related quality of life (HRQL). The overall CCQ consists of 10 items that are scored from 0 to 6. The final score is the sum of all items divided by 10. Higher scores indicate a worse health status.
Assessment of Depression | 6 months
  Assessment of the potential effect of self-management intervention on depression using Beck Depression Inventory, 2nd edition (BDI).The Beck Depression Inventory (BDI) is a 21-item self-reporting questionnaire for evaluating the severity of depression in normal and psychiatric populations.Scores range from zero to 60. Higher total scores indicate more severe depressive symptoms.
Assessement of Anxiety | 6 months
  Assessment of the potential effect of self-management intervention on anxiety using Beck Anxiety Inventory (BAI). The BAI is a rating scale used to evaluate the severity of anxiety symptoms. The total score ranges from 0 to 63, with higher scores indicating more severe anxiety symptoms.
Assessement of Patient education | 6 months
  Assessment of the potential effect of self-management intervention on patient education, using Health Education Impact Questionnaire (HeiQ), for evaluating the training intervention. Responses to 40 items are marked on a 4-point Likert scale, using the endpoints "strongly disagree/strongly agree". A higher score indicates stronger skills in the management of the chronic condition, except in the emotional distress dimension, which is negatively scored.
Assessment of Functional status | 6 months
  Assessment of the potential effect of self-management intervention on functional status using Modified Medical Research Council Dyspnea Scale (mMRC) to assess dyspnea.The mMRC breathlessness scale ranges from grade 0 to 4. Higher scores indicate greater severity of breathlessness.
Assessement of Patient education | 6 months
  Assessment of the potential effect of self-management intervention on patient education, using Health Literacy Questionnaire (HLQ), assessing literacy.The full HLQ provides nine individual scores based on an average of the items within each of the nine scales. Higher values indicate greater understanding or ability.

CONTACTS AND LOCATIONS:
Overall Officials: Ioanna Tsiligianni, Study Chair — University of Crete, Greece
Locations (1):
- University of Crete, Heraklion, Greece

IPD SHARING:
Plan to Share IPD: No